CLINICAL TRIAL: NCT04515238
Title: A Prospective, Open-label, Multicenter Phase-II Trial to Evaluate the Efficacy and Safety of a Sequential Regimen of Bendamustine Followed by Obinutuzumab (GA101), Zanubrutinib (BGB-3111) and Venetoclax (ABT-199) in Patients With Relapsed/Refractory CLL (CLL2-BZAG Protocol)
Brief Title: Sequential Regimen of Bendamustine Followed by Obinutuzumab (GA101), Zanubrutinib (BGB-3111) and Venetoclax (ABT-199) in Patients With Relapsed/Refractory CLL
Acronym: CLL2-BZAG
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL2-BZAG; 2022-502201-16-00 (EU CTIS Number); 2018-003270-27 (EudraCT Number)
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Chronic Lymphoid Leukemia
Keywords: CLL
MeSH Terms: conditions — Leukemia, B-Cell | interventions — Bendamustine Hydrochloride; obinutuzumab; zanubrutinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BZAG (Experimental): Debulking: 2 debulking cycles (q 28d) of bendamustine will be administered unless the patient has a contraindication or a debulking is not clinically indicated
  Induction: 6 cycles (q 28d) of Obinutuzumab + Zanubrutinib + Venetoclax
  Maintenance: max. 8 cycles (q 84d) of Obinutuzumab + Zanubrutinib + Venetoclax
  Maintenance treatment will be continued until (whichever occurs first):
  * 12 weeks (approx. 3 months) after confirmation of achievement of a CR/CRi and MRD negativity
  * maintenance cycle 8
  * progression of CLL or start of a subsequent therapy unacceptable toxicity
  Interventions: Drug: Bendamustine; Biological: Obinutuzumab; Biological: Zanubrutinib; Biological: Venetoclax

INTERVENTIONS:
Drug: Bendamustine — Debulking: Cycles 1-2: d1+2 - 70mg/m² i.v.
  Other Names: Treanda; Bendeka
Biological: Obinutuzumab — Induction: Cycle 1: d1 - 100 mg, d1 (or d2) - 900 mg, d8 + d15 - 1000 mg i.v.; Cycle 2 - 6: 1000 mg, d1 i.v.
  Maintenance: Cycle 1 - 8: 1000 mg, d1 i.v.
  Other Names: GA101; Gazyvaro
Biological: Zanubrutinib — Induction: Cycle 1: --; Cycles 2 - 6: d1-28: 2 x 160mg p.o.
  Maintenance: Cycle 1 - 8: d1-84: 2 x 160mg p.o
  Other Names: BGB-3111
Biological: Venetoclax — Induction: Cycles 1 + 2: --; Cycle 3: d1-7: 20mg, d8-14: 50mg, d15-21: 100mg, d22-28: 200mg p.o.; Cycle 4 - 6: d1-28: 400 mg p.o.
  Maintenance: Cycle 1 - 8: d1-84: 400 mg p.o.
  Other Names: ABT-199; Venclyxto

SUMMARY:
CLL2-BZAG is a prospective, open-label, multicenter phase-II trial to evaluate the efficacy and safety of a sequential regimen of bendamustine followed by obinutuzumab (GA101), zanubrutinib (BGB-3111) and venetoclax (ABT-199) in patients with relapsed/refractory CLL.

DETAILED DESCRIPTION:
In the CLL2-BZAG trial will be included a total of 40 patients with relapsed or refractory CLL in need of treatment. This trial will evaluate a debulking with two cycles bendamustine (only for patients with a high tumor load), followed by an induction and maintenance treatment with obinutuzumab, zanubrutinib and venetoclax in patients with relapsed/refractory CLL. Thus, this trial combines one established (chemotherapy) and three novel, synergistic (antibody, Bruton's tyrosine kinase(BTK)-inhibitor and Bcl-2 antagonist) principles of action in order to achieve deep and long lasting remissions with a short duration of treatment. Additionally, this trial has an extensive accompanying scientific program aiming at a better understanding of the kinetics of response and clonal evolution of CLL.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed/refractory CLL in need of treatment according to International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria

   In case of a recent previous treatment, patients must have recovered from acute toxicities and treatment regimen must be stopped within the following time periods before start of the study treatment in the CLL2-BZAG trial:
   * chemotherapy ≥ 28 days
   * antibody treatment ≥ 14 days
   * kinase inhibitors, BCL2-antagonists or immunomodulatory agents ≥ 3 days
   * corticosteroids may be applied until the start of the BZAG-regimen, these have to be reduced to an equivalent of ≤ 20mg prednisolone per day during treatment Please note: Patients with a progression during previous treatment with venetoclax, ibrutinib or another BTK inhibitor, as well as patients with a known resistance mutation (e.g. BTK-/PLCg2) are excluded from study participation. However, patients who progressed after termination of treatment with venetoclax, ibrutinib, other BTK inhibitors and/or obinutuzumab or who stopped treatment due to intolerance to ibrutinib are eligible for participation.
2. Adequate renal function, as indicated by a creatinine clearance ≥30ml/min calculated according to the modified formula of Cockcroft and Gault or directly measured with 24 hr. urine collection
3. Adequate hematologic function as indicated by a neutrophil count ≥ 1.0 x 109/L, a hemoglobin value ≥8.0 g/dL and a platelet count ≥ 25 x 109/L, unless directly attributable to the patient´s CLL (e.g. bone marrow infiltration), in this case, platelet count should be ≥ 10 × 109/L.
4. Adequate liver function as indicated by a total bilirubin ≤2x, AST/ALT ≤2.5x the institutional ULN value, unless directly attributable to the patient's CLL or to Gilbert's Syndrome
5. Negative serological testing for hepatitis B (HBsAg negative and anti-HBc negative, patients positive for anti-HBc may be included if PCR for Hepatitis B Virus (HBV) DNA is negative and HBV-DNA PCR is performed every 4 weeks until one year after last dosage of GA101 (obinutuzumab) or until the last dose of zanubrutinib, whichever occurs later), negative testing for hepatitis-C RNA and negative HIV test within 6 weeks prior to registration
6. Age ≥ 18 years
7. Eastern Cooperative Oncology Group Performance Status (ECOG) 0 - 2, ECOG 3 is only permitted if related to CLL (e.g. due to anemia or severe constitutional symptoms)
8. Life expectancy ≥ 6 months
9. Ability and willingness to provide written informed consent and to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

1. (Suspicion of) transformation of CLL (i.e. Richter's transformation, pro-lymphocytic leukemia) or central nervous system (CNS) involvement
2. Progression during previous treatment with venetoclax, ibrutinib or another BTK inhibitor, and/or presence of known mutations associated with resistance to therapy, e.g. Bruton´s Tyrosine Kinase and Phospholipase C Gamma 2 (PLCg2)
3. Confirmed progressive multifocal leukoencephalopathy (PML)
4. Malignancies other than CLL currently requiring systemic therapies
5. Uncontrolled infection requiring systemic treatment
6. Any comorbidity or organ system impairment rated with a Cumulative Illness Rating Scale (CIRS) score of 4, excluding the eyes/ears/nose/throat/larynx organ system or any other life-threatening illness, medical condition or organ system dysfunction that - in the investigator´s opinion - could compromise the patients safety or interfere with the absorption or metabolism of the study drugs (e.g, inability to swallow tablets or impaired resorption in the gastrointestinal tract)
7. Significantly increased risk of bleeding according to the investigator´s evaluation, e.g. due known bleeding diathesis (e.g. von-Willebrandt´s disease or hemophilia), major surgical procedure ≤ 4 weeks or stroke/intracranial hemorrhage ≤ 6 months.
8. Requirement of therapy with strong CYP3A4 inhibitors/inducers or anticoagulant with phenprocoumon (marcumar) or other vitamin K-antagonists
9. Use of investigational agents ≤ 28 days prior to start of study treatment, however, kinase inhibitors, BCL2-antagonists and antibody treatment are allowed in accordance with inclusion criterion number 1 (see above).
10. Known hypersensitivity to obinutuzumab (GA101), venetoclax (ABT-199), zanubrutinib (BGB-3111) or any of the excipients Please note: Patients with a known hypersensitivity to bendamustine are allowed to participate but will not receive a debulking with bendamustine
11. Pregnant women and nursing mothers (a negative pregnancy test is required for all women of childbearing potential within 7 days before start of treatment)
12. Fertile men or women of childbearing potential unless:

    * surgically sterile or ≥ 2 years after the onset of menopause, or
    * willing to use two methods of reliable contraception including one highly effective (Pearl Index <1) and one additional effective (barrier) method during study treatment and for 18 months after end of study treatment.
13. Vaccination with a live vaccine ≤ 28 days prior to registration
14. Legal incapacity
15. Prisoners or subjects who are institutionalized by regulatory or court order
16. Persons who are in dependence to the sponsor or an investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Negativity rate of minimal residual disease (MRD) in peripheral blood (PB) measured by multi-color flow cytometry | At final restaging (RE): 12 weeks after the start of the last induction cycle
  MRD negativity is defined as less than one (1) CLL-cell among 10,000 leukocytes analyzed [0.01%]. The MRD negativity rate is defined as the proportion of patients having achieved MRD negativity based on the full analysis set (FAS).

SECONDARY OUTCOMES:
Overall response rate (ORR) | At final restaging (RE): 12 weeks after the start of the last induction cycle
  Proportion of patients having achieved a complete response (CR), a CR with incomplete recovery of the bone marrow (CRi), or a partial response (PR) as best response.
CR / CRi rate | At final restaging (RE): 12 weeks after the start of the last induction cycle
  Proportion of patients having achieved a CR or CRi as best response (= number of patients with best response CR or CRi divided by the number of the FAS)
MRD in PB measured by 4-color flow cytometry at different times to guide the duration of maintenance therapy and for the assessment of the kinetics of response to the different treatment phases | From date of screening until the end of follow-up, up to 55 month
  MRD negativity is defined as less than one (1) CLL-cell among 10,000 leukocytes analyzed [0.01%], i.e. < 10-4. MRD values will be categorized into negative (<10-4) and positive (≥10-4)
Safety: Adverse events (AE), serious adverse events (SAE) and adverse events of particular/special interest (AEPI/AESI) | Up to 55 months after first dose of study drug
  Type, frequency, severity and relationship to study treatment.of AEs, SAEs and AEPIs/AESIs

CONTACTS AND LOCATIONS:
Overall Officials: Paula Cramer, Dr. med., Principal Investigator — German CLL Study Group
Locations (11):
- Germany (11):
  - Hamatologische/Onkologische Gemeinschaftspraxis, Augsburg
  - Universitätsklinik Köln, Cologne
  - Onkologische Schwerpunktpraxis, Esslingen am Neckar
  - Evangelische Krankenhaus Hamm, Hamm
  - Universitaetskliniken des Saarlandes, Homburg
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - KH Kliniken Maria Hilf, Mönchengladbach
  - Klinikum Rechts der Isar - Technische Universitaet Muenchen, Munich
  - Stauferklinikum Schwaebisch-Gmuend, Mutlangen
  - Universitätsklinik Ulm, Ulm
  - Hämatologisch Onkologische Schwerpunktpraxis, Würzburg

REFERENCES:
- [Derived] Furstenau M, Robrecht S, Schneider C, Tausch E, Giza A, Ritgen M, Bittenbring J, Hebart H, Schottker B, Illert AL, Graeven U, Stoltefuss A, Heinrich B, Eckert R, Fink A, Stumpf J, Fischer K, Al-Sawaf O, Simon F, Kleinert F, Weiss J, Kreuzer KA, Schilhabel A, Bruggemann M, Langerbeins P, Stilgenbauer S, Eichhorst B, Hallek M, Cramer P. MRD-guided zanubrutinib, venetoclax, and obinutuzumab in relapsed CLL: primary end point analysis from the CLL2-BZAG trial. Blood. 2025 Mar 20;145(12):1282-1292. doi: 10.1182/blood.2024026685. PMID 39883943
- See also: Click here for more information about this study: CLL2-BZAG (German CLL Study Group) — https://www.dcllsg.com/cll2-bzag/
- See also: MRD-guided zanubrutinib, venetoclax, and obinutuzumab in relapsed CLL: primary end point analysis from the CLL2-BZAG trial. Blood. 2025 Mar 20;145(12):1282-1292. doi: 10.1182/blood.2024026685. PMID: 39883943. — https://pubmed.ncbi.nlm.nih.gov/39883943/